CLINICAL TRIAL: NCT00027365
Title: A Phase I Safety and Immunogenicity Trial of a Combination Vaccine (NefTat and gp120w61d) Formulated With AS02A (GlaxoSmithKline Biologicals) Given Intramuscularly in HIV-1 Uninfected Adult Participants
Brief Title: An Investigational Combination Vaccine Given to People Who Are Not Infected With HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 041; 10196 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2001-12-04; First posted 2001-12-05 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; Injections, Intramuscular; HIV Antibodies; HIV-1; HIV Envelope Protein gp120; Gene Products, tat; AIDS Vaccines; Neutralization Tests; Vaccines, Combined; AIDS Seronegativity; Gene Products, nef
MeSH Terms: conditions — HIV Infections | interventions — Vaccines, Combined

INTERVENTIONS:
Biological: Combination Vaccine (NefTat and gp120W61D) Formulated with AS02A
Biological: NefTat
Drug: AS02A Adjuvant
Biological: gp120W61D

SUMMARY:
The purpose of this study is to see if the investigational vaccines NefTat and gp120w61d are safe and tolerable in humans and to see how the immune system responds to the vaccines.

There have been advances in the treatment and prevention of HIV, but the spread of HIV/AIDS is getting worse. HIV/AIDS is the main infectious cause of death in the world. A vaccine to prevent HIV disease is the best way to try to deal with this situation. Several vaccine products have been tested, but only 2 are still in trial. There is a need for a new product.

DETAILED DESCRIPTION:
Despite recent advances in the treatment and prevention of HIV disease, the epidemic is worsening throughout most of the world. HIV/AIDS is the leading cause of death in sub-Saharan Africa and the leading infectious cause of death in the world. An effective and inexpensive vaccine to prevent HIV disease remains as the best option to try to deal with this expanding epidemic. A number of vaccine products have been tested; however, only 2 have progressed to a Phase III trial, underscoring the need for new vaccine strategies.

Prior to study entry, participants have their risk status for HIV infection determined by a series of questions. Further eligibility is determined by results of physical exam, laboratory tests, and further questions. Blood is drawn on each study visit. Participants are assigned randomly to 1 of 4 study groups:

Group I: NefTat or placebo. Groups II, III, and IV: NefTat and gp120 or placebo. Each group receives a different concentration of gp120.

All immunizations are admixed with AS02A adjuvant. Vaccinations are administered intramuscularly at 3 time points (entry, 1 month, and 3 months). Product safety and immunogenicity are performed at designated time points; participants have about 11 clinic visits.

ELIGIBILITY:
Inclusion Criteria

Participants may be eligible for this study if they:

* Are between 18 and 60 years of age.
* Are in good general health and meet laboratory test requirements.
* Have a CD4 count of 400 or more cells/mm3.
* Agree to use at least 1 of the following methods of contraception for at least 21 days before enrollment until the last protocol visit: condoms (male or female) with or without a spermicide, diaphragm or cervical cap with spermicide, IUD, or hormonal-based therapy (applies to women who are able to have children).
* Have access to a participating site and are willing to have follow-up for the entire study (12 months).
* Answer questions about their understanding of the study.
* Do not have hepatitis B or C.
* Are HIV-uninfected.

Exclusion Criteria

Participants may not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Have recently received a vaccine.
* Have used experimental agents within 30 days before enrollment.
* Have received HIV vaccines or placebo in a previous HIV vaccine study.
* Have received blood products 120 days before HIV screening.
* Have received immunoglobulin (antibodies) 60 days before HIV screening.
* Have serious reactions to vaccines.
* Have problems with their immune system.
* Have cancer.
* Have used drugs that affect the immune system within the past 6 months.
* Have diabetes.
* Have a thyroid disease.
* Have unstable asthma.
* Are taking anti-tuberculosis drugs.
* Have seizures.
* Have a bleeding disorder.
* Have had their spleen removed.
* Have angioedema (a certain type of body tissue swelling).
* Have active syphilis.
* Have high blood pressure (unless controlled by medication).
* Have mental or emotional problems that make them unsuitable for the study.
* Have any medical, mental, or social condition; job responsibilities; or other responsibility that, in the opinion of the doctor, would interfere with the study.
* Have reactions to components of the vaccines.
* Are at high risk for contracting HIV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84
Dates: Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Evans, Study Chair
Locations (15):
- United States (15):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Johns Hopkins Bloomberg School of Public Health,Ctr for Immunization Research, Project SAVE-Baltimore, Baltimore, Maryland
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Fenway Community Health Clinical Research Site (FCHCRS), Boston, Massachusetts
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - NY Blood Ctr./Union Square CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - NY Blood Ctr./Bronx CRS, The Bronx, New York
  - Miriam Hospital's HVTU, Providence, Rhode Island
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - Infectious Diseases Physicians, Inc., Annandale, Virginia
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Result] Vaine M, Wang S, Liu Q, Arthos J, Montefiori D, Goepfert P, McElrath MJ, Lu S. Profiles of human serum antibody responses elicited by three leading HIV vaccines focusing on the induction of Env-specific antibodies. PLoS One. 2010 Nov 9;5(11):e13916. doi: 10.1371/journal.pone.0013916. PMID 21085486